CLINICAL TRIAL: NCT01479127
Title: An Open-Label, Single-Arm, Baseline-Controlled, Multicenter Study to Explore the Safety, Tolerability, Pharmacokinetics, and Efficacy of ABT-SLV187 in Subjects With Advanced Parkinson's Disease
Brief Title: Study of Safety, Tolerability, Pharmacokinetics, and Efficacy of ABT-SLV187 in Subjects With Advanced Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Abbott Japan Co.,Ltd (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-925
Record Dates: First submitted 2011-09-26; First posted 2011-11-24 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Advanced Parkinson's Disease
Keywords: Levodopa-carbidopa intestinal gel; Advanced Parkinson's disease; Severe motor fluctuations; Dyskinesia
MeSH Terms: conditions — Dyskinesias | interventions — carbidopa, levodopa drug combination; Carbidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levodopa-carbidopa intestinal gel (Experimental): Following a 28-day Run-in Period where participants are switched from prior anti-PD medications to monotherapy with an oral 100 mg levodopa/10 mg carbidopa tablet (optimized every 3rd hour during waking hours), participants receive ABT-SLV187 (levodopa-carbidopa intestinal gel), administered over 16 hours a day with an infusion pump directly into the proximal jejunum by an NJ tube, for 3 weeks.
  The individually-adjusted infusion dose (composed of the morning dose, the continuous maintenance dose, and the extra dose) is optimized by the Investigator for each participant during the study based on the participant's symptoms.
  Interventions: Drug: ABT-SLV187; Drug: Oral Levodopa/Carbidopa; Device: Infusion Pump: CADD-Legacy® 1400 Pump; Device: NJ-Tube: Silicon ED Tube; Device: Adaptor: Hakko Adaptor

INTERVENTIONS:
Drug: ABT-SLV187
  Other Names: DUOPA™ (carbidopa and levodopa Enteral Suspension); DUODOPA®; Levodopa-carbidopa intestinal gel (LCIG)
Drug: Oral Levodopa/Carbidopa — Tablet; contains 100 mg levodopa and 10 mg carbidopa
Device: Infusion Pump: CADD-Legacy® 1400 Pump — General infusion pump, manufactured by Smiths Medical (US)
Device: NJ-Tube: Silicon ED Tube — Device used to deliver nutrition/drug to stomach/intestine or to aspirate stomach fluid, manufactured by Create Medic Co., Ltd. (Japan)
Device: Adaptor: Hakko Adaptor — Accessory set for fluid infusion set, consisting of caps, connectors and adapters, etc, manufactured by Hakko Medical (Japan)

SUMMARY:
To explore the safety, tolerability, pharmacokinetics and efficacy of ABT-SLV187 in advanced Parkinson's disease (PD) patients with severe motor complications. The complications of medical devices for the naso-jejunum (NJ) infusion system of ABT-SLV187 will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD according to the United Kingdom Parkinson's Disease Society (UKPDS) Brain Bank criteria
* PD stage corresponds to 4 or 5 in the 'off' state according to the modified Hoehn & Yahr (H & Y) classification of disease severity
* Levodopa-responsive subjects demonstrate some identifiable 'ON response' established by observation by Investigator and demonstrate severe motor fluctuations in spite of individually optimized treatment and where therapy options are indicated

Exclusion Criteria:

* Diagnosis is unclear or a suspicion of other parkinsonian syndromes exists such as secondary parkinsonism
* Undergone surgery for the treatment of PD
* Contraindications to levodopa
* Subjects with any neurological deficit that may interfere with the study assessments

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yukihiro Kumamoto, MS, Study Director — AbbVie Japan Co., Ltd

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Levodopa-carbidopa Intestinal Gel: Following a 28-day Run-in Period where participants are switched from prior anti-Parkinson's disease (PD) medications to monotherapy with an oral 100 mg levodopa/10 mg carbidopa tablet (optimized every 3rd hour during waking hours), participants receive ABT-SLV187 (levodopa-carbidopa intestinal gel [LCIG]), administered over 16 hours a day with an infusion pump directly into the proximal jejunum by a naso-jejunum (NJ) tube, for 3 weeks.
  The individually-adjusted infusion dose (composed of the morning dose, the continuous maintenance dose, and the extra dose) is optimized by the Investigator for each participant during the study based on the participant's symptoms.
Period: Overall Study
Arm/Group | Levodopa-carbidopa Intestinal Gel
Started | 8 (started oral study drug (full safety sample))
Started LCIG | 6
Completed | 5
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: full safety sample
Groups:
- Levodopa-carbidopa Intestinal Gel: Following a 28-day Run-in Period where participants are switched from prior anti-PD medications to monotherapy with an oral 100 mg levodopa/10 mg carbidopa tablet (optimized every 3rd hour during waking hours), participants receive ABT-SLV187 (levodopa-carbidopa intestinal gel), administered over 16 hours a day with an infusion pump directly into the proximal jejunum by a naso-jejunum (NJ) tube, for 3 weeks.
  The individually-adjusted infusion dose (composed of the morning dose, the continuous maintenance dose, and the extra dose) is optimized by the Investigator for each participant during the study based on the participant's symptoms.
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (6.19)
Age, Customized [Number; unit: participants]
  < 65 years | 4
  >/= 65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), and AEs Leading to Discontinuation During the Run-in Period
Description: AE: any untoward medical occurrence in a participant that does not necessarily have a causal relationship with this treatment. SAE: an event that results in the death of a subject, is life threatening, results in hospitalization or prolongation of hospitalization, is a congenital anomaly, results in persistent or significant disability/incapacity, or other important medical event. Severity was rated as mild, moderate, or severe. AEs of special interest included: device-associated gastrointestinal disorders; cardiovascular fatalities; aspiration including aspiration pneumonia; a diagnosis of peripheral polyneuropathy (axonal, demyelinating or mixed type); possible symptoms of peripheral polyneuropathy; clinically significant weight loss. 'AEs at least possibly related' are defined as those that were assessed by investigator as probably related or possibly related.
Time Frame: During the Run-in period (up to approximately 28 days)
Population: Full safety sample: participants who had at least one dose of oral levodopa-carbidopa study drug in the Run-in Period.
Measure: Number; unit: participants
Groups:
- Oral Levodopa/Carbidopa Tablet: During a 28-day Run-in Period, participants are switched from prior anti-PD medications to monotherapy with an oral 100 mg levodopa/10 mg carbidopa tablet (optimized every 3rd hour during waking hours)
Arm/Group | Oral Levodopa/Carbidopa Tablet
Number analyzed (Participants) | 8
participants
  AE | 7
  AE at least possibly related to study drug/device | 5
  Severe AE | 0
  SAE | 0
  AE leading to discontinuation of study drug | 1
  SAE at least possibly drug or drug device-related | 0
  AE of special interest | 0
  AE caused by study drug | 5
  AE caused by devices | NA — Not applicable to Run-in Period.
  AE caused by NJ tube insertion | NA — Not applicable to Run-in Period.
  Fatal AE | 0

2. Primary Outcome: Number of Participants With AEs, SAEs, and AEs Leading to Discontinuation During the ABT-SLV187 Treatment Period
Description: as for outcome 1
Time Frame: From NJ placement to end of ABT-SLV187 Treatment Period (Day 21) +30 days
Population: ABT-SLV187 safety sample: participants who had at least one dose of the ABT-SLV187 study medication after the baseline assessment.
Measure: Number; unit: participants
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 6
participants
  AE | 4
  AE at least possibly related to study drug/device | 3
  Severe AE | 1
  SAE | 1
  AE leading to discontinuation of study drug | 1
  SAE at least possiby drug or drug device-related | 1
  AE of special interest | 2
  AE caused by study drug | 3
  AE caused by devices | 0
  AE caused by NJ tube insertion | 1
  Fatal AE | 0

3. Primary Outcome: Number of Participants With Potentially Clinically Significant (PCS) Hematology Results During the ABT-SLV187 Treatment Period
Description: M=male, F=female, MCV=mean corpuscular volume, MCH=mean corpuscular hemoglobin, MCHC=mean corpuscular hemoglobin concentration.
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 6
participants
  Low PCS Hematocrit [%]: 39.8 M / 33.4 F | 3
  High PCS Hematocrit [%]: 51.8 M / 44.9 F | 0
  Low PCS Hemoglobin [g/dL]: 13.5 M / 11.3 F | 3
  High PCS Hemoglobin [g/dL]: 17.6 M / 15.2 F | 0
  Low PCS RBC Count [*10^4/µL]: 427 M / 376 F | 3
  High PCS RBC Count [*10^4/µL]: 570 M / 500 F | 0
  Low PCS WBC Count [/µL]: 3900 M / 3500 F | 1
  High PCS WBC Count [/µL]: 9800 M / 9100 F | 0
  Low PCS Neutrophils [%]: 40.0 | 0
  High PCS Neutrophils [%]: 74.0 | 0
  Low PCS Lymphocytes [%]: 18.0 | 0
  High PCS Lymphocytes [%]: 59.0 | 0
  Low PCS Monocytes [%]: 0.0 | 0
  High PCS Monocytes [%]: 8.0 | 1
  Low PCS Basophils [%]: 0.0 | 0
  High PCS Basophils [%]: 2.0 | 0
  Low PCS Eosinophils [%]: 0.0 | 0
  High PCS Eosinophils [%]: 6.0 | 0
  Low PCS Platelet count [*10^4/µL]: 13.1 M / 13.0 F | 0
  High PCS Platelet count [*10^4/µL]: 36.2 M/ 36.9 F | 1
  Low PCS MCV [FL]: 82.7 M / 79.0 F | 0
  High PCS MCV [FL]: 101.6 M / 100.0 F | 0
  Low PCS MCH [Pg]: 28 M / 26.3 F | 0
  High PCS MCH [Pg]: 34.6 M / 34.3 F | 0
  Low PCS MCHC [%]: 31.6 M / 30.7 F | 1
  High PCS MCHC [%]: 36.6 M / 36.6 F | 0

4. Primary Outcome: Number of Participants With PCS Blood Biochemistry Results During the ABT-SLV187 Treatment Period
Description: M=male, F=female, γ-GTP=gamma-glutamyl transpeptidase.
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 6
participants
  Low PCS Blood urea nitrogen [mg/dL]: 6 | 0
  High PCS Blood urea nitrogen [mg/dL]: 20 | 1
  Low Creatinine [mg/dL]: 0.61 M / 0.47 F | 2
  High Creatinine [mg/dL]: 1.04 M / 0.79 F | 0
  Low PCS Total bilirubin [mg/dL]: 0.2 | 0
  High PCS Total bilirubin [mg/dL]: 1.0 | 0
  Low PCS Alanine aminotransferase [U/L]: 5 | 0
  High PCS Alanine aminotransferase [U/L]: 40 | 0
  Low PCS Aspartate aminotransferase [U/L]: 10 | 1
  High PCS Aspartate aminotransferase [U/L]: 40 | 0
  Low PCS Alkaline phosphatase [U/L]: 115 | 0
  High PCS Alkaline phosphatase [U/L]: 359 | 1
  Low PCS γ-GTP [U/L]: 0 | 0
  High PCS γ-GTP [U/L]: 70 M / 30 F | 0
  Low PCS Sodium [mEq/L]: 136 | 1
  High PCS Sodium [mEq/L]: 147 | 0
  Low PCS Potassium [mEq/L]: 3.6 | 0
  High PCS Potassium [mEq/L]: 5.0 | 0
  Low PCS Calcium [mg/dL]: 8.7 | 3
  High PCS Calcium [mg/dL]: 10.1 | 0
  Low PCS Chloride [mEq/L]: 98 | 1
  High PCS Chloride [mEq/L]: 109 | 0
  Low PCS Magnesium [mg/dL]: 1.8 | 0
  High PCS Magnesium [mg/dL]: 2.6 | 1
  Low PCS Inorganic Phosphors [mg/dL]: 2.4 | 0
  High PCS Inorganic Phosphors [mg/dL]: 4.3 | 1
  Low PCS Uric acid [mg/dL]: 3.7 M / 2.5 F | 2
  High PCS Uric acid [mg/dL]: 7 M / 7.0 F | 0
  Low PCS Total cholesterol [mg/dL]: 150 | 0
  High PCS Total cholesterol [mg/dL]: 219 | 2
  Low PCS Total protein [g/dL]: 6.7 | 5
  High PCS Total protein [g/dL]: 8.3 | 0
  Low PCS Albumin [g/dL]: 4.0 | 3
  High PCS Albumin [g/dL]: 5.0 | 0
  Low PCS Glucose [mg/dL]: 70 | 0
  High PCS Glucose [mg/dL]: 109 | 1
  Low PCS Triglycerides [mg/dL]: 50 | 1
  High PCS Triglycerides [mg/dL]: 149 | 0
  Low PCS Creatine kinase [U/L]: 57 M / 32 F | 1
  High PCS Creatine kinase [U/L]: 197 M / 180 F | 3
  Low PCS Bicarbonate [mEq/L]: 22 | 0
  High PCS Bicarbonate [mEq/L]: 29 | 0
  Low PCS Lactate dehydrogenase [U/L]: 115 | 0
  High PCS Lactate dehydrogenase [U/L]: 245 | 1

5. Primary Outcome: Number of Participants With PCS Values in Special Laboratory Parameters During the ABT-SLV187 Treatment Period
Description: M=male, F=female
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 6
participants
  Low PCS Vitamin B6 pyridoxamine [ng/mL]: </= 0.6 | 0
  Low PCS Vitamin B6 pyridoxal [ng/mL]: 6.0 M/4.0 F | 4
  High PCS Vitamin B6 pyridoxal [ng/mL]: 40 M / 19 F | 1
  Low PCS Vitamin B6 pyridoxine [ng/mL]: </= 3.0 | 0
  Low PCS Vitamin B12 [pg/mL]: 180 | 1
  High PCS Vitamin B12 [pg/mL]: 914 | 0
  Low PCS Homocysteine [nmol/mL]: 3.7 | 0
  High PCS Homocysteine [nmol/mL]: 13.5 | 4
  Low PCS Folic acid [ng/mL]: < 3.1 | 1

6. Secondary Outcome: Mean Change From Baseline to the End of Treatment in Percentage of Ratings in the "OFF" and "Dyskinesia" States on the TRS I and the "Normal," "OFF," and "Dyskinesia" States on the TRS II
Description: Participants were video recorded a total of 10 times for 1 to 2 minutes every 60 minutes while performing a standardized sequence of motor tasks: rest, finger taps, rapid alternating movement of hands, arising from chair and gait, including confirmation of postural stability. Based on these video recordings, a Video Evaluation Committee consisting of 3 neurologists individually evaluated the following Video Assessment and TRS under blinded conditions: Finger Taps, Rapid Alternating Movement of Hands, Arising from Chair, Gait, Body Bradykinesia and Hypokinesia, Dyskinesia for TRS I, with the addition of Tremor at Rest and Postural Stability for TRS II. The average of the 3 neurologists' evaluations was calculated as a percentage of ratings in the "Normal" state (ie, "mild OFF" to "ON with mild dyskinesia"), the "Off" state ("moderate OFF" to "severe OFF"), and the "Dyskinesia" state ("ON with moderate dyskinesia" to "ON with severe dyskinesia") on the TRS I or II.
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: Full Analysis Set: participants who had data for baseline and at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: percentage of ratings
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5
percentage of ratings
  TRS I "OFF" state | -15.33 (13.04)
  TRS I "Dyskinesia" state | 0.00 (4.71)
  TRS II "Normal" state | 14.67 (18.65)
  TRS II "OFF" state | -15.33 (18.65)
  TRS II "Dyskinesia" state | 0.67 (1.49)
Statistical Analysis 1: Comparison: Levodopa-carbidopa Intestinal Gel; TRS I "OFF" state; Test type: Superiority or Other; p = 0.058, Paired t-test
Statistical Analysis 2: Comparison: Levodopa-carbidopa Intestinal Gel; TRS I "Dyskinesia" state; Test type: Superiority or Other; p = 1.000, Paired t-test
Statistical Analysis 3: Comparison: Levodopa-carbidopa Intestinal Gel; TRS II "Normal" state; Test type: Superiority or Other; p = 0.153, Paired t-test
Statistical Analysis 4: Comparison: Levodopa-carbidopa Intestinal Gel; TRS II "OFF" state; Test type: Superiority or Other; p = 0.140, Paired t-test
Statistical Analysis 5: Comparison: Levodopa-carbidopa Intestinal Gel; TRS II "Dyskinesia" state; Test type: Superiority or Other; p = 0.374, Paired t-test

7. Secondary Outcome: Change From Baseline to the End of Treatment in Parkinson's Disease Diary Assessment
Description: For each half hour period during 3 consecutive days prior to each assessment of the diary, participants (and/or their caregivers) entered into a diary whether they were asleep, in the ON motor state or in the OFF motor state in the following 5 grades: asleep, OFF, ON (no dyskinesia [D]), ON with non-troublesome dyskinesia (NTD), ON with troublesome dyskinesia (TD). ON time is when PD symptoms are well controlled by the drug. OFF time is when PD symptoms are not adequately controlled by the drug. Dyskinetic time is time with involuntary muscle movement. The ON or OFF times were calculated as the average of 3 daily times from the diaries. w/o = without, w/ = with
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: Full Analysis Set: participants who had data for baseline and at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5
hours
  Daily OFF time | -1.02 (3.73)
  Daily ON time w/o D + time w/ NTD | 0.76 (3.61)
  Daily ON time w/o D + time w/ NTD + time w/ TD | 1.02 (3.73)
Statistical Analysis 1: Comparison: Levodopa-carbidopa Intestinal Gel; Test type: Superiority or Other; p = 0.574, Paired t-test
Statistical Analysis 2: Comparison: Levodopa-carbidopa Intestinal Gel; ON time w/o D + time with NTD; Test type: Superiority or Other; p = 0.661, Paired t-test
Statistical Analysis 3: Comparison: Levodopa-carbidopa Intestinal Gel; ON time w/o D + time with NTD + time w/ TD; Test type: Superiority or Other; p = 0.574, Paired t-test

8. Secondary Outcome: Baseline and Endpoint (End of Treatment) Video Scoring of Unified Parkinson's Disease Rating Scale (UPDRS) Items and Dyskinesia
Description: Participants were video recorded a total of 10 times for 1 to 2 minutes every 60 minutes while performing a standardized sequence of motor tasks. Based on these video recordings, a Video Evaluation Committee consisting of 3 neurologists individually evaluated the video under blinded conditions using the following assessments: Tremor at Rest (UPDRS item #20), Finger Taps (UPDRS #23), Rapid Alternating Movement of Hands (UPDRS #25), Arising from Chair (UPDRS #27), Gait (UPDRS #29), Postural Stability (UPDRS #30), Body Bradykinesia and Hypokinesia (UPDRS #31), and Dyskinesia (evaluated with the Goetz Dyskinesia Rating Scale). The UPDRS score is the sum of the answers to individual questions, each of which are measured on a 5-point scale (0-4), with higher scores associated with more disability. The Goetz Dyskinesia Rating Scale is a 5-point scale of the severity of dyskinesias, from 0 (absent) to 4 (violent dyskinesias).
Time Frame: Baseline (Day -1), Endpoint (Day 21)
Population: Full Analysis Set: participants who had data for baseline and at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5
units on a scale
  Tremor at rest, Baseline | 0.00 (0.00)
  Tremor at rest, Endpoint | 0.00 (0.00)
  Finger taps, Baseline | 0.40 (0.55)
  Finger taps, Endpoint | 0.40 (0.55)
  Rapid alternating movement of hands, Baseline | 1.00 (0.00)
  Rapid alternating movement of hands, Endpoint | 0.60 (0.55)
  Arising from chair, Baseline | 0.10 (0.22)
  Arising from chair, Endpoint | 0.00 (0.00)
  Gait, Baseline | 0.60 (0.55)
  Gait, Endpoint | 0.60 (0.55)
  Postural stability, Baseline | 1.60 (0.55)
  Postural stability, Endpoint | 1.10 (0.89)
  Body bradykinesia and hypokinesia, Baseline | 1.00 (0.00)
  Body bradykinesia and hypokinesia, Endpoint | 0.80 (0.27)
  Dyskinesia, Baseline | 0.40 (0.55)
  Dyskinesia, Baseline | 0.90 (0.55)
Statistical Analysis 1: Comparison: Levodopa-carbidopa Intestinal Gel; Rapid alternating movement of hands; Test type: Superiority or Other; p = 0.500, Wilcoxon one-sample test
Statistical Analysis 2: Comparison: Levodopa-carbidopa Intestinal Gel; Arising from chair; Test type: Superiority or Other; p = 1.000, Wilcoxon one-sample test
Statistical Analysis 3: Comparison: Levodopa-carbidopa Intestinal Gel; Postural stability; Test type: Superiority or Other; p = 0.250, Wilcoxon one-sample test
Statistical Analysis 4: Comparison: Levodopa-carbidopa Intestinal Gel; Body bradykinesia and hypokinesia; Test type: Superiority or Other; p = 0.500, Wilcoxon one-sample test
Statistical Analysis 5: Comparison: Levodopa-carbidopa Intestinal Gel; Dyskinesia; Test type: Superiority or Other; p = 0.250, Wilcoxon one-sample test

9. Secondary Outcome: Mean Change From Baseline to the End of Treatment in UPDRS Total Scores and Subscores
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The total score is the sum of the responses to the 31 questions (44 answers) that comprise Parts I-III of the scale. The total score ranges from 0-176, with 176 representing the worst (total) disability, and 0 no disability. The Part I Score is the sum of the answers to the 4 questions related to Mentation, Behavior and Mood, and ranges from 0-16. The Part II score is the sum of the answers to the 13 questions related to Activities of Daily Living, and ranges from 0-52. The Part III score is the sum of the 27 answers related to Motor Examination, and ranges from 0-108. The Part IV Score is the sum of the answers to the 11 questions related to Complications of Therapy, and ranges from 0-23. The Part IV dyskinesia subscore ranges from 0-12. For each part of the UPDRS, higher scores are associated with more disability.
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: Full Analysis Set: participants who had data for baseline and at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5
units on a scale
  Total score | -0.60 (7.70)
  Part I | 0.20 (0.45)
  Part II | 0.60 (4.93)
  Part II (Off-time) | -2.20 (6.54)
  Part III | -1.40 (4.56)
  Part IV subscore of dyskinesia | 2.20 (2.39)
Statistical Analysis 1: Comparison: Levodopa-carbidopa Intestinal Gel; Total score; Test type: Superiority or Other; p = 0.870, Paired t-test
Statistical Analysis 2: Comparison: Levodopa-carbidopa Intestinal Gel; Part I; Test type: Superiority or Other; p = 0.374, Paired t-test
Statistical Analysis 3: Comparison: Levodopa-carbidopa Intestinal Gel; Part II; Test type: Superiority or Other; p = 0.799, Paired t-test
Statistical Analysis 4: Comparison: Levodopa-carbidopa Intestinal Gel; Part II (Off-time); Test type: Superiority or Other; p = 0.493, Paired t-test
Statistical Analysis 5: Comparison: Levodopa-carbidopa Intestinal Gel; Part III; Test type: Superiority or Other; p = 0.530, Paired t-test
Statistical Analysis 6: Comparison: Levodopa-carbidopa Intestinal Gel; Part IV sub-score of dyskinesia; Test type: Superiority or Other; p = 0.108, Paired t-test

10. Secondary Outcome: Change From Baseline to the End of Treatment in the Japanese Version of Parkinson's Disease Questionnaire 39 (PDQ-39) Total Score and Domain Scores
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients, including Mobility, Activities of Daily Living, Emotional Well-being, Stigma, Social Support, Cognition, Communication, and Bodily Discomfort, as well as a Summary Index Total Score. Scores for each are on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: Full Analysis Set: participants who had data for baseline and at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5
units on a scale
  Total score | 1.26 (5.48)
  Domain: Mobility | 10.00 (20.16)
  Domain: Activities of daily living | -0.83 (14.25)
  Domain: Emotional well-being | -8.33 (12.84)
  Domain: Stigma | 1.25 (10.27)
  Domain: Social support | -5.00 (6.85)
  Domain: Cognition | -5.00 (13.55)
  Domain: Communication | 1.67 (20.75)
  Domain: Bodily discomfort | 8.33 (30.62)
Statistical Analysis 1: Comparison: Levodopa-carbidopa Intestinal Gel; Total score; Test type: Superiority or Other; p = 0.636, Paired t-test
Statistical Analysis 2: Comparison: Levodopa-carbidopa Intestinal Gel; Domain: Mobility; Test type: Superiority or Other; p = 0.329, Paired t-test
Statistical Analysis 3: Comparison: Levodopa-carbidopa Intestinal Gel; Domain: Activities of daily living; Test type: Superiority or Other; p = 0.902, Paired t-test
Statistical Analysis 4: Comparison: Levodopa-carbidopa Intestinal Gel; Domain: Emotional well-being; Test type: Superiority or Other; p = 0.220, Paired t-test
Statistical Analysis 5: Comparison: Levodopa-carbidopa Intestinal Gel; Domain: Stigma; Test type: Superiority or Other; p = 0.799, Paired t-test
Statistical Analysis 6: Comparison: Levodopa-carbidopa Intestinal Gel; Domain: Social support; Test type: Superiority or Other; p = 0.178, Paired t-test
Statistical Analysis 7: Comparison: Levodopa-carbidopa Intestinal Gel; Domain: Cognition; Test type: Superiority or Other; p = 0.456, Paired t-test
Statistical Analysis 8: Comparison: Levodopa-carbidopa Intestinal Gel; Domain: Communication; Test type: Superiority or Other; p = 0.866, Paired t-test
Statistical Analysis 9: Comparison: Levodopa-carbidopa Intestinal Gel; Domain: Bodily discomfort; Test type: Superiority or Other; p = 0.576, Paired t-test

11. Secondary Outcome: Modified Hoehn and Yahr Staging at Baseline and End of Treatment
Description: Participant's ON and OFF states staged according to the Modified Hoehn and Yahr criteria, an 8-point scale for staging: 0, No signs of disease; 1, Unilateral disease; 1.5, Unilateral plus axial involvement; 2, Bilateral disease; 2.5, Mild bilateral disease; 3, Mild to moderate bilateral disease; 4, Severe disability; and 5, Wheelchair bound or bedridden unless aided. ON time is when PD symptoms are well controlled by the drug. OFF time is when PD symptoms are not adequately controlled by the drug.
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: Full Analysis Set: participants who had data for baseline and at least one post-baseline efficacy measurement.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5
units on a scale
  ON state staging, Baseline | 2.5 [2.5 to 3]
  ON state staging, Endpoint | 3.0 [2 to 3]
  OFF state staging, Baseline | 4.0 [4 to 4]
  OFF state staging, Endpoint | 4.0 [2 to 4]
Statistical Analysis 1: Comparison: Levodopa-carbidopa Intestinal Gel; "On" state staging; Test type: Superiority or Other; p = 1.000, Wilcoxon one-sample test
Statistical Analysis 2: Comparison: Levodopa-carbidopa Intestinal Gel; "Off" state staging; Test type: Superiority or Other; p = 1.000, Wilcoxon one-sample test

12. Secondary Outcome: Schwab and England Activities of Daily Living Scale at Baseline and End of Treatment
Description: The Schwab and England scale was used to rate the subject's activities of daily living by recording the percentage score, ranging between being completely independent (100%) and totally dependent (10%).
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: Full Analysis Set: participants who had data for baseline and at least one post-baseline efficacy measurement.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5
units on a scale
  Baseline | 80.0 [50 to 80]
  Endpoint | 80.0 [70 to 90]
Statistical Analysis 1: Comparison: Levodopa-carbidopa Intestinal Gel; Test type: Superiority or Other; p = 0.125, Wilcoxon one-sample test

13. Secondary Outcome: Clinical Global Impression - Severity (CGI-S) Score at Baseline and Clinical Global Impression - Improvement (CGI-I) Score at Baseline and End of Treatment
Description: The CGI-S is a global assessment by the Investigator of current symptomatology and impact of illness on functioning. The ratings of the CGI-S are as follows: normal, borderline ill, mildly ill, moderately ill, markedly ill, severely ill, and among the most extremely ill. The CGI-I is a global assessment by the Investigator of the change in clinical status since the start of treatment. The CGI-I ratings are as follows: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse.
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: Full Analysis Set: participants who had data for baseline and at least one post-baseline efficacy measurement.
Measure: Number; unit: participants
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5
participants
  CGI-S, Baseline: Normal | 0
  CGI-S, Baseline: Borderline ill | 0
  CGI-S, Baseline: Mildly ill | 0
  CGI-S, Baseline: Moderately ill | 2
  CGI-S, Baseline: Markedly ill | 3
  CGI-S, Baseline: Severely ill | 0
  CGI-S, Baseline: Among the most extremely ill | 0
  CGI-S, Endpoint: Normal | 1
  CGI-S, Endpoint: Borderline ill | 0
  CGI-S, Endpoint: Mildly ill | 0
  CGI-S, Endpoint: Moderately ill | 3
  CGI-S, Endpoint: Markedly ill | 1
  CGI-S, Endpoint: Severely ill | 0
  CGI-S, Endpoint: Among the most extremely ill | 0
  CGI-I: Very much improved | 1
  CGI-I: Much improved | 3
  CGI-I: Minimally improved | 1
  CGI-I: No change | 0
  CGI-I: Minimally worse | 0
  CGI-I: Much worse | 0
  CGI-I: Very much worse | 0

14. Primary Outcome: Number of Participants With Potentially Clinically Significant Urinalysis Results During the ABT-SLV187 Treatment Period
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 6
participants
  Low PCS Specific gravity: 1.002 | 0
  High PCS Specific gravity: 1.030 | 0
  Low PCS pH: 4.5 | 0
  High PCS pH: 8.0 | 1
  High PCS Protein: > trace | 0
  High PCS Glucose: > trace | 0
  High PCS Occult blood: > negative | 0
  High PCS Ketone: > negative | 0

15. Primary Outcome: Number of Participants With Potentially Clinically Significant (PCS) Vital Signs Results During the ABT-SLV187 Treatment Period
Description: ↓=decrease, ↑=increase, BL=baseline, temp.=temperature, SBP=systolic blood pressure, Sup.=supine, Sta.=standing, DBP=diastolic blood pressure.
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 6
participants
  Low PCS Weight [kg]: ≥7% ↓ from BL | 0
  High PCS Weight [kg]: ≥7% ↑ from BL | 0
  High PCS Body temp. [⁰C]: ≥38.8 and ≥1.1 ↑ from BL | 0
  Low PCS SBP Sup. [mmHg]: ≤90 and >30 ↓ from BL | 0
  High PCS SBP Sup. [mmHg]: ≥180 and >40 ↑ from BL | 0
  Low PCS SBP Sta. [mmHg]: ≤90 and >30 ↓ from BL | 1
  High PCS SBP Sta. [mmHg]: ≥180 and >40 ↑ from BL | 0
  Low PCS SBP Orthostatic [mmHg]: ↓ of ≥30 in SBP | 1
  Low PCS DBP Sup. [mmHg]: ≤50 and >30 ↓ from BL | 0
  High PCS DBP Sup. [mmHg]: ≥105 and >30 ↑ from BL | 0
  Low PCS DBP Sta. [mmHg]: ≤50 and >30 ↓ from BL | 0
  High PCS DBP Sta. [mmHg]: ≥105 and >30 ↑ from BL | 0
  Low PCS DBP Orthostatic [mmHg]: ↓ of ≥20 in DBP | 1
  Pulse rate [bpm]: ≤50 and >30 ↓ from BL | 0
  Pulse rate [bpm]: ≥120 and >30 ↑ from BL | 0

16. Primary Outcome: Number of Participants With Potentially Clinically Significant 12-lead Electrocardiogram (ECG) Results During the ABT-SLV187 Treatment Period
Description: High potentially clinically significant Bazett's heart rate-corrected QT interval (QTcB) values were: 450 msec for males / 470 msec for females.
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 6
participants | 0

17. Primary Outcome: Mean Change From Baseline to the End of Treatment in Percentage of Ratings in the "Normal" State on the Treatment Response Scale (TRS) I
Description: Participants were video recorded a total of 10 times for 1 to 2 minutes every 60 minutes while performing a standardized sequence of motor tasks: rest, finger taps, rapid alternating movement of hands, arising from chair and gait, including confirmation of postural stability. Based on these video recordings, a Video Evaluation Committee consisting of 3 neurologists individually evaluated the following Video Assessment and Treatment Response Scale (TRS) under blinded conditions: Finger Taps, Rapid Alternating Movement of Hands, Arising from Chair, Gait, Body Bradykinesia and Hypokinesia, Dyskinesia. The average of the neurologists' evaluations was calculated as a percentage of ratings in the "Normal" state (ie, "mild OFF" to "ON with mild dyskinesia") on the TRS I (total 10 assessments per day).
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: Full Analysis Set: participants who had data for baseline and at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: percentage of ratings
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5
percentage of ratings | 15.33 (14.26)
Statistical Analysis 1: Comparison: Levodopa-carbidopa Intestinal Gel; Test type: Superiority or Other; p = 0.074, Paired t-test

18. Secondary Outcome: Time to Reach Peak Plasma Concentration (Tmax) After Administration of Oral Levodopa/Carbidopa (L/C) Tablets and Intra-jejunal Administration of ABT-SLV187
Description: Tmax of levodopa, carbidopa, and its metabolite 3-O-methyldopa (3-OMD) after administration of oral L/C tablets and intra-jejunal administration of ABT-SLV187.
Time Frame: Baseline (Day -1): pre-dose; 15, 30, 45, 60 mins post-morning dose; every 30 mins thereafter for 12 hrs. Day 21: pre-dose; 15, 30, 45, 60 mins post-infusion; every 30 mins from hrs 1 to 12 post-infusion; every 2 hrs from 12 to 16 hrs post-infusion.
Population: Pharmacokinetic (PK) sample: participants who completed PK assessments in both the oral L/C and ABT-SLV187 Treatment Periods.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Oral Levodopa-carbidopa Tablets: A 28-day Run-in Period where participants are switched from prior anti-PD medications to monotherapy with an oral 100 mg levodopa/10 mg carbidopa tablet (optimized every 3rd hour during waking hours).
- Levodopa-carbidopa Intestinal Gel: Participants receive ABT-SLV187 (levodopa-carbidopa intestinal gel), administered over 16 hours a day with an infusion pump directly into the proximal jejunum by an NJ tube, for 3 weeks.
  The individually-adjusted infusion dose (composed of the morning dose, the continuous maintenance dose, and the extra dose) is optimized by the Investigator for each participant during the study based on the participant's symptoms.
Arm/Group | Oral Levodopa-carbidopa Tablets | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5 | 5
hours
  Levodopa | 3.0 (3.5) | 1.0 (0.50)
  Carbidopa | 7.8 (2.8) | 4.5 (4.2)
  3-OMD | 11 (0.76) | 11 (0.79)

19. Secondary Outcome: Peak Plasma Concentration (Cmax), Average Plasma Concentration (Cavg), Trough Plasma Concentration (Cmin), and Cmin Within 2 and 12 Hours (Cmin [2-12 Hours]) After Administration of Oral L/C Tablets and Intra-jejunal Administration of ABT-SLV187
Description: Cmax, Cavg, Cmin, and Cmin (2-12 hours) of levodopa, carbidopa, and 3-OMD after administration of the oral L/C tablets (Day -1) and intra-jejunal administration of ABT-SLV187 (Day 21). Cmin values for levodopa and carbidopa during the 16 hours of infusion were observed either at time 0 or 15 min after start of the infusion and were a result of drug washout prior to establishment of infusion.
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: PK sample: participants who completed PK assessments in both the oral L/C and ABT-SLV187 Treatment Periods.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Oral Levodopa-carbidopa Tablets | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5 | 5
µg/mL
  Cmax: Levodopa | 5.96 (0.77) | 4.38 (1.15)
  Cmax: Carbidopa | 0.128 (0.03) | 0.273 (0.07)
  Cmax: 3-OMD | 9.27 (2.17) | 11.7 (1.25)
  Cavg: Levodopa | 2.37 (0.26) | 2.87 (0.66)
  Cavg: Carbidopa | 0.079 (0.02) | 0.172 (0.04)
  Cavg: 3-OMD | 7.36 (1.93) | 9.80 (1.23)
  Cmin: Levodopa | 0.268 (0.43) | 0.061 (0.03)
  Cmin: Carbidopa | 0.014 (0.02) | 0.016 (0.01)
  Cmin: 3-OMD | 5.67 (1.60) | 7.78 (0.63)
  Cmin (2-12 hours): Levodopa | 0.734 (0.43) | 2.38 (0.77)
  Cmin (2-12 hours):Carbidopa | 0.050 (0.02) | 0.130 (0.04)
  Cmin (2-12 hours): 3-OMD | 5.72 (1.53) | 8.14 (0.94)

20. Secondary Outcome: The Area Under the Concentrations-time Curve From 0 to 12 and 0 to 16 Hours (AUC0-12, AUC0-16) After Administration of Oral L/C Tablets and Intra-jejunal Administration of ABT-SLV187
Description: AUC0-12 and AUC0-16 of levodopa, carbidopa, and 3-OMD after administration of the oral L/C tablets (Day -1) and intra-jejunal administration of ABT-SLV187 (Day 21).
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: PK sample: participants who completed PK assessments in both the oral L/C and ABT-SLV187 Treatment Periods.
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Oral Levodopa-carbidopa Tablets | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5 | 5
µg*h/mL
  AUC0-12: Levodopa | 28.4 (3.08) | 34.4 (7.95)
  AUC0-12: Carbidopa | 0.94 (0.18) | 2.07 (0.52)
  AUC0-12: 3-OMD | 88.3 (23.1) | 118 (14.7)
  AUC0-16: Levodopa | NA (NA) — AUC0-16 for oral levodopa-carbidopa tablets was not assessed. | 46.7 (10.7)
  AUC0-16: Carbidopa | NA (NA) — AUC0-16 for oral levodopa-carbidopa tablets was not assessed. | 2.80 (0.666)
  AUC0-16: 3-OMD | NA (NA) — AUC0-16 for oral levodopa-carbidopa tablets was not assessed. | 165 (21.2)

21. Secondary Outcome: AUC0-12/Dose0-12, AUC0-16/Dose0-16 After Administration of Oral L/C Tablets and Intra-jejunal Administration of ABT-SLV187
Description: AUC0-12/Dose0-12 of levodopa, carbidopa, and 3-OMD after administration of the oral L/C tablets (Day -1) and intra-jejunal administration of ABT-SLV187 (Day 21). AUC0-16/Dose0-16 of levodopa, carbidopa, and 3-OMD after administration of intra-jejunal administration of ABT-SLV187 (Day 21).
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: PK sample: participants who completed PK assessments in both the oral L/C and ABT-SLV187 Treatment Periods.
Measure: Mean (Standard Deviation); unit: µg*h/mL/mg
Arm/Group | Oral Levodopa-carbidopa Tablets | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5 | 5
µg*h/mL/mg
  AUC0-12/Dose0-12: Levodopa | 0.036 (0.008) | 0.032 (0.006)
  AUC0-12/Dose0-12: Carbidopa | 0.012 (0.003) | 0.008 (0.001)
  AUC0-12/Dose0-12: 3-OMD | 0.112 (0.029) | 0.113 (0.022)
  AUC0-16/Dose0-16: Levodopa | NA (NA) — AUC0-16/Dose0-16 not applicable after administration of the oral L/C tablets (Day -1). | 0.035 (0.007)
  AUC0-16/Dose0-16: Carbidopa | NA (NA) — AUC0-16/Dose0-16 not applicable after administration of the oral L/C tablets (Day -1). | 0.008 (0.001)
  AUC0-16/Dose0-16: 3-OMD | NA (NA) — AUC0-16/Dose0-16 not applicable after administration of the oral L/C tablets (Day -1). | 0.125 (0.025)

22. Secondary Outcome: Degree of Fluctuation (2-12 Hours) After Administration of Oral L/C Tablets and Intra-jejunal Administration of ABT-SLV187
Description: Degree of Fluctuation (calculated as [Cmax - Cmin] / Cavg)) of levodopa, carbidopa, and 3-OMD after administration of the oral L/C tablets (Day -1) and intra-jejunal administration of ABT-SLV187 (Day 21).
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: PK sample: participants who completed PK assessments in both the oral L/C and ABT-SLV187 Treatment Periods.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Oral Levodopa-carbidopa Tablets | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5 | 5
ratio
  Levodopa | 2.1 (0.59) | 0.38 (0.16)
  Carbidopa | 0.97 (0.20) | 0.78 (0.25)
  3-OMD | 0.48 (0.10) | 0.35 (0.07)

23. Secondary Outcome: Ratio of Metabolite 3-OMD to Levodopa (M/P [AUC0-12]) After Administration of Oral L/C Tablets and Intra-jejunal Administration of ABT-SLV187
Description: M/P (AUC0-12) after administration of the oral L/C tablets (Day -1) and intra-jejunal administration of ABT-SLV187 (Day 21).
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: PK sample: participants who completed PK assessments in both the oral L/C and ABT-SLV187 Treatment Periods.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Oral Levodopa-carbidopa Tablets | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 5 | 5
ratio | 3.11 (0.71) | 3.53 (0.70)

24. Secondary Outcome: Number of Participants With Product Quality Complaints (PQC) During the ABT-SLV187 Treatment Period
Time Frame: Baseline (Day -1), End of ABT-SLV187 Treatment Period (Day 21)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Levodopa-carbidopa Intestinal Gel
Number analyzed (Participants) | 6
participants
  Any PQC | 2
  Any PQC related to an AE | 0
  Any serious PQC | 0
  Any PQC leading to discontinuation of study drug | 0
  Any PQC by pump | 0
  Any PQC by NJ-tube insertion | 2
  Any PQC by adapter | 0
  Any PQC by cassettes | 1
  Without any PQCs | 4

ADVERSE EVENTS:
Time Frame: AEs: from the time of first study drug administration in the Run-in Period to 30 days following completion or discontinuation of study drug administration (up to 79 days). SAEs from the time of Screening (up to 93 days).
Arm/Group | Oral Levodopa-carbidopa Tablets | Levodopa-carbidopa Intestinal Gel
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/6
Other Adverse Events (participants affected / at risk) | 7/8 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Levodopa-carbidopa Tablets (N=8) | Levodopa-carbidopa Intestinal Gel (N=6)
Delusion (Psychiatric disorders) | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 1
Somatic hallucination (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Levodopa-carbidopa Tablets (N=8) | Levodopa-carbidopa Intestinal Gel (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Intentional medical device removal by patient (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 1
Otitis externa (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
ON and OFF phenomenon (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 0
Rapid eye movements sleep abnormal (Psychiatric disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.